CLINICAL TRIAL: NCT02826876
Title: Local Analgesia in Laparoscopic Surgery
Brief Title: The Efficacy of Surgical Site Treatment With Ropivacaine in Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Farraj Moaad, Dr, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0196-15-NHR
Record Dates: First submitted 2016-06-22; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Pain
Keywords: Laparoscopic surgery
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine (Placebo Comparator): Topical use of Ropivacaine
  Interventions: Drug: Topical use; Other: laparoscopic repair of inguinal hernia; Other: laparoscopic bariatric surgery
- Placebo (Placebo Comparator): Topical use of placebo
  Interventions: Drug: Topical use; Other: laparoscopic repair of inguinal hernia; Other: laparoscopic bariatric surgery

INTERVENTIONS:
Drug: Topical use — Topical use of Ropivacaine in laparoscopic surgery
  Other Names: Ropivacaine; Placebo
Other: laparoscopic repair of inguinal hernia — intra-operative treatment with ropivacaine Vs placebo in laparoscopic repair of inguinal hernia
Other: laparoscopic bariatric surgery — intra-operative treatment with ropivacaine Vs placebo in laparoscopic bariatric surgery

SUMMARY:
Using local analgesia in laparoscopic surgery in order to reduce pain and to reduce the use of narcotic drugs.

DETAILED DESCRIPTION:
At the end of laparoscopic surgery the investigators will spray ropivacaine in the surgical site; and later the investigators will monitor pain intensity and use of analgesic drugs

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic bariatric surgery
* Laparoscopic inguinal hernia surgery

Exclusion Criteria:

* Cardiac arrythmias
* Active ischemic heart disease
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Pain scale as measured by pain scale questionnaire | 1 Week
  post operative pain intensity will be assisted by VAS(visual analog pain scale) scale at fixed times after surgery

SECONDARY OUTCOMES:
Reducing use of narcotics according to nurse records | 1 Week
  patients will be treated by standard analgetic protocol, the records of analgetic drugs will be collected during patients hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Moaad H Farraj, Dr, Principal Investigator — Galilee Medical Center
Locations (1):
- Naharia Medical Center, Nahariya, Israel